CLINICAL TRIAL: NCT03324763
Title: Study of the Performances of a Fast Diagnosis Immunochromatographic Test for the Detection of Helicobacter Pylori (H. Pylori) Antigens in Child Stool
Brief Title: Performances of a Fast Test for the Detection of Helicobacter Pylori Antigens in Child Stool
Acronym: DISPOSE
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Collaborators: Hôpital Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: RT-10
Record Dates: First submitted 2017-10-25; First posted 2017-10-30 (Actual); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Helicobacter Pylori Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool of children
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- stool sampling
  Interventions: Other: stool sampling

INTERVENTIONS:
Other: stool sampling — A stool sample will be collected to perform the H. pylori antigen test

SUMMARY:
The diagnostic tests used to detect Helicobacter pylori (H. pylori) infection are either direct and invasive, as in culture, histology and the rapid urease test (RUT) or noninvasive, such as serology, the 13C-Urea breathe test or the stool antigen test. However, there is no single reference method to detect the H. pylori infection reliably and accurately. The specificity of gastric biopsy cultures is 100%, but the sensitivity is lower. Histology and RUT provide excellent diagnostic accuracy, but the detection of H. pylori is decreased in cases of bleeding peptic ulcers or gastric atrophy. Therefore, it is recommended that at least two tests should agree when defining the H. pylori infection in children. Quantitative real-time polymerase chain reaction (qPCR)-based methods have been shown to be the most reliable for H. pylori detection in adults and in children. In children, the reference method for H. pylori infection detection is invasive, namely upper digestive endoscopy with gastric biopsy for histology, culture, RUT and qPCR. A noninvasive alternative to detect H. pylori antigen in stools could use a quick one-step immuno-chromatographic technique.

The aim of this study was to assess the performance of a new quick, noninvasive, one-step immuno-chromatographic, stool antigen test (ALERE Inc, Jouy-en-Josas, France) for the detection of H. pylori infection in children.

ELIGIBILITY:
Inclusion Criteria:

* Children <18 years old
* All children undergoing a high digestive endoscopy with per-endoscopic gastric biopsies.
* Informed consent of parents and children

Exclusion Criteria:

* Children having received an antibiotic treatment 4 weeks before inclusion
* Children having received Proton pump inhibitors 2 weeks before inclusion
* Children having received Bismuth salts 2 weeks before inclusion

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with various digestive symptoms suggesting upper gastrointestinal tract disease consulting at Saint Antoine paediatric clinic, Saint Vincent de Paul Hospital, Lille-France.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2014-03-19 (Actual); Primary Completion 2015-10-07 (Actual); Study Completion 2015-10-07 (Actual)

PRIMARY OUTCOMES:
Performance of a new quick, noninvasive, one-step immuno-chromatographic, stool antigen test France) for the detection of H. pylori infection in children | Baseline
  The performances of the diagnostic test will be assess by considering the reference test as Gold Standard

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Saint Vincent de Paul, Lille, Hauts-de-France, France

IPD SHARING:
Plan to Share IPD: No